CLINICAL TRIAL: NCT03862612
Title: Efficacy of Serratus Anterior Plane (SAP) Block Versus Erector Spinae Plane (ESP) Block for Quality of Recovery After Video Assisted Thoracic Surgery : A Randomised Control Trial
Brief Title: Efficacy of SAP Block Versus ESP Block in VATS Surgery
Acronym: ESPvSAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mater Misericordiae University Hospital (Other)
Responsible Party: Principal Investigator, Dylan Finnerty, Principal Investigator, Mater Misericordiae University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ESPverusSAP
Record Dates: First submitted 2019-02-28; First posted 2019-03-05 (Actual); Last update posted 2020-05-04 (Actual); Status verified 2020-04

CONDITIONS: Regional Anesthesia Morbidity
MeSH Terms: interventions — Anesthesia, Conduction

STUDY DESIGN:
Intervention Model Description: randomised control trial one group receives Serratus Anterior Plane Block the other receives Erector Spinae Plane Block
Who Masked: Participant, Care Provider, Investigator
Masking Description: Blocks will be administered after induction of General Anesthesia so participants will be blinded to which intervention they have had.
  Study investigators will not be aware as to what group the participant belongs to when assessing the patient post operative period
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector Spinae Plane Block (Active Comparator): This group will receive an Erector Spinae Plane Block under ultrasound guidance while under General Anaesthesia
  Interventions: Procedure: regional anaesthesia with Levobupivicaine 0.25% 30mls with two methods either erector spinae plane block or serratus anterior plane block
- Serratus Anterior Plane Block (Experimental): This group will receive a Serratus Anterior Plane Block under ultrasound guidance while under General Anesthesia
  Interventions: Procedure: regional anaesthesia with Levobupivicaine 0.25% 30mls with two methods either erector spinae plane block or serratus anterior plane block

INTERVENTIONS:
Procedure: regional anaesthesia with Levobupivicaine 0.25% 30mls with two methods either erector spinae plane block or serratus anterior plane block — Erector Spinae Plane Block will be compared to the Serratus Anterior Plane Block in patients undergoing Video assissted thoracic surgery

SUMMARY:
During VATS (Video assisted thoracic surgery) small incisions are made in the patient's chest through which a camera and instruments are inserted to allow a lung operation to be performed. Often patients experience a substantial amount of pain and difficult recovery after this type of operation. Anaesthesiologists sometimes use "Regional Anaesthesia" to minimise the pain and help patient recovery after the operation. This involves injecting local anaesthesia into the nerves around the chest wall to effectively numb that part of the chest. There is a variety of different locations on the chest wall where the local anaesthetic can be deposited and no study has measured whether one technique is better than the other in terms of improving patients' recovery experience. Our study compares two new techniques for Regional Anaesthesia after this type of surgery. Participants will be randomly assigned (like tossing a coin) to receive either a SAP (Serratus Anterior Plane) or ESP (Erector Spinae Plane) Block. Both techniques are described within last five years, but have never been compared for chest surgery

DETAILED DESCRIPTION:
The Serratus Anterior Plane (SAP) Block has been claimed to be a safer, technically less demanding alternative to paravertebral block and thoracic epidural in the management of post operative VATS associated pain . Recently, another new block, the Erector Spinae Block (ESP Block) has been described for use in thoracic wall surgery. It has also been claimed to be easier to perform than these more traditional methods of regional anaesthesia. No study to date has compared ESP to SAP blocks in terms of efficacy of post operative analgesia after VATS surgery. Furthermore, patient-centres outcome studies now demand that researchers evaluate more than acute pain in the early postoperative period: A 15-parameter Quality of Recovery score (QoR-15) has been recommended as the optimum tool to evaluate overall patient-centres measures of recovery after surgery, including pain. This study will test the hypothesis that patients receiving ESP Block have higher QoR-15 scores and better post operative analgesia in comparison with patients receiving SAP Block after VATS surgery.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female participants providing written informed consent,
* ASA grade 1- 4,
* aged over 18
* undergoing a VATS procedure under General Anaesthesia

Exclusion Criteria:

* Absence of informed written consent,
* pre existing infection at block site,-
* severe coagulopathy,
* allergy to local anaesthesia,
* pre existing neurological deficit,
* previous history of opiate abuse,
* pre existing chronic pain condition,
* pre-existing dementia [because of need to co-operate in completing QoR-15 score day after surgery].

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-06-05 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2020-04-02 (Actual)

PRIMARY OUTCOMES:
the patient centred QoR-15 score among ESB and SAP block patients; | 1 year
  A 15-parameter Quality of Recovery score (QoR-15) has been recommended as the optimum tool to evaluate overall patient-centres measures of recovery after surgery, including pain. It is a questionnaire that is given to patients to do post operatively and is scored from 0 to 150 where 150 indicates that the patient has a had an excellent recovery

SECONDARY OUTCOMES:
Area under the Verbal Rating Scale (VRS) pain score versus time (24 hr post-op | 24 hours post op
  Verbal Rating Scale pain score is measured from 0 to 10 where 0 is no pain and 10 is severe pain
. VRS pain scores at 1 hr, 12 hr, 24 hr postop | 24 hours post op
  0-10 where 10 equals severe pain and 0 is no pain
time to administration of first rescue analgesia after the block | 24hours post op
documentation of adverse events : hypotension, pruritus, nausea and vomiting | 24 hours post op

CONTACTS AND LOCATIONS:
Overall Officials: Donal Buggy, Principal Investigator — Professor of Anaesthesia and Perioperative Medicine
Locations (1):
- Mater Misericordiae University Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Finnerty DT, McMahon A, McNamara JR, Hartigan SD, Griffin M, Buggy DJ. Comparing erector spinae plane block with serratus anterior plane block for minimally invasive thoracic surgery: a randomised clinical trial. Br J Anaesth. 2020 Nov;125(5):802-810. doi: 10.1016/j.bja.2020.06.020. Epub 2020 Jul 11. PMID 32660716